CLINICAL TRIAL: NCT00662168
Title: An Investigation of Eight Reported Cases of Small Intestinal Carcinoid Carcinoma in Multiple Family Members
Brief Title: An Investigation of Small Intestinal Carcinoid Carcinoma in Families
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rutgers University (Other)
Responsible Party: Nancy Gardner, PhD. Assistant Professor, Rutgers University
Other Study IDs: 08-151
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Carcinoid Carcinoma
Keywords: carcinoid; familial; Collect and describe information about the medical and environmental factors associated with each cases of carcinoid carcinoma; Develop a genogram representing the family cancer history of cases of Carcinoid.
MeSH Terms: conditions — Carcinoid Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation: Individuals with a diagnosis of carcinoid carcinoma

SUMMARY:
This proposed pilot study is to conduct detailed interviews into the medical, environmental, and family histories The second phase of this study project is to and to collect blood specimen to obtain DNA. The Blood specimen and DNA will be processed by the Rutgers University Cell and DNA Repository (RUCDR) and stored for a second phase of this pilot. The purpose is to rule out Familial Multiple Endocrine Neoplasia (MEN 1), and succinate dehydrogenase complex, subunit D (SDHD), gene inactivation thought to be associated with different types of carcinoid cancer.

DETAILED DESCRIPTION:
There have not been any studies published which specifically describe the medical, environmental, and genetic factors in carcinoid tumors cases that have carcinoid in family members. While rare, with an incidence of four per 100, 000, carcinoid represents the most frequent malignancy affecting the small intestine. Because nearly half (49%) of the cases of gastrointestinal carcinoid tumors have hepatic metastasis at diagnosis, identification of the risk factors associated with carcinoid has the potential to increase early diagnosis and cure. Carcinoid tumors are thought to occur spontaneously and not associated with an inherited genetic abnormality that would increase a family member's risk for developing carcinoid cancer. There is a known inherited genetic abnormality that is associated with bronchial carcinoid tumors but only less than 10%. Gastrointestinal carcinoid tumors are not thought to be associated with a inherited genetic abnormality. There have been several small studies that have examined gastrointestinal carcinoid in multiple family members. It remains uncertain if these cases of carcinoid in multiple family members are characteristic of a heritable or environmental etiology. Most carcinoid cancer is not inherited; however, less than 10% of neuroendocrine carcinoid cancer is thought to be due to a change (called a "mutation") in a gene inherited from a parent. There are several genes that are suspected to be associated with carcinoid cancer, two of interest in this study is the Multiple Endocrine Neoplasia Type1 (MEN1), and succinate dehydrogenase complex, subunit D (SDHD) genes.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years
2. History of biopsy confirmed small intestinal carcinoid tumor
3. English speaking
4. Mentally and emotionally capable of answering questions
5. Willing and available for study participation
6. At least one first-degree family member with carcinoid tumor

Exclusion Criteria:

1. If you are under the age of 18 years,
2. If you have any mental or memory impairments
3. If you are unable to understand the information in the informed consent document.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with carcinoid cancer that report to have a family member also with carcinoid tumor
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
identification of carcinoid in multiple family members | lifetime history

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Gardner, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University College of Nursing, Newark, New Jersey, United States